CLINICAL TRIAL: NCT06371872
Title: French Cohort of Patients With Rotator Cuff Lesions: Changes in Shoulder Function and Quality of Life at 1, 2, 5, 8 and 10 Years, According to Their Care
Brief Title: French Cohort of Patients With Rotator Cuff Lesions
Acronym: PRO-CUFF
Status: Not yet recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2024-A00173-44
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with rotator cuff injuries: Patients will be recruited during their first consultation for treatment of a rotator cuff injury. Patients will then be contacted by telephone or e-mail every year to monitor the progress of their disease and their treatment.
  Patients will be asked to complete self-questionnaires assessing shoulder function, quality of life and satisfaction. These questionnaires will be accessible via a secure website.
  Interventions: Procedure: total transfixing injury to the rotator cuff

INTERVENTIONS:
Procedure: total transfixing injury to the rotator cuff — develop an appropriate prescription strategy with a view to improving patients' quality of life in the short, medium and long term in this condition

SUMMARY:
The purpose of this study is to identify, at 5 years, the clinical and therapeutic factors associated with improvement in shoulder functionality and quality of life in patients with transfixing (total) rotator cuff injuries undergoing treatment.

DETAILED DESCRIPTION:
This is a non-interventional, prospective, longitudinal, multicentre cohort study.

The research procedure involves recruiting patients during their first consultation for the management of a rotator cuff injury. Patients will then be contacted by telephone or e-mail every year to monitor the progress of their disease and their treatment. Patients will be asked to complete self-questionnaires assessing shoulder function, quality of life and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age.
* Patient with a transfixing (total) rotator cuff lesion confirmed by imaging.
* A patient who has been informed and has expressed no oral objection to taking part in the research.
* Patient affiliated to or benefiting from a social security scheme.

Exclusion Criteria:

* Patients over 75 years of age.
* Patients with a history of shoulder surgery.
* Patients unable to receive emails and/or answer online questionnaires.
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients recruited during their first consultation for the management of a rotator cuff injury.
Sampling Method: Non-Probability Sample
Enrollment: 519 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | 5 years
  Improved shoulder function (evolution of SPADI score, composed of a pain sub-score and a shoulder mobility sub-score ≥ 13 points compared with inclusion)
European quality of life scale - EQ5D | 5 years
  Improved quality of life (change in EQ5D score ≥ 0.1 points from baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Maussins-Nollet, Paris, France